CLINICAL TRIAL: NCT07360340
Title: Methotrexate Therapy and High-Resolution CT Chest and Spirometry Test Findings in Egyptian Patients With Rheumatoid Arthritis.
Brief Title: Methotrexate Therapy and High-Resolution CT Chest and Spirometry Test Findings in Patients With Rheumatoid Arthritis.
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: FMASU Ms 778/2022
Record Dates: First submitted 2026-01-01; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-12

CONDITIONS: Methohexitone Pulmonary Adverse Reaction
Keywords: Methotrexate Therapy,; CT Chest; Spirometry Test; Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group A 25 patients on methotrexate therapy, Group B 25 patients not on methotrexate: Group A: - 25 RA patients treated with MTX only +/- low dose steroid. Group B: - 25 MTX naive RA patients (treated with DMARDs other than MTX) +/- low dose steroid.

SUMMARY:
ABSTRACT Background: Rheumatoid arthritis (RA) is characterized by symmetrical erosive synovitis and progressive disability, often complicated by extra-articular manifestations especially in seropositive patients, among them, lung involvement is common, and it can include a wide spectrum of disorders, ranging from airways, pleural disease, bronchiectasis, lung nodules, to infection.

Aim of the Work: The aim of this study is to assess HRCT Chest and spirometry test findings in RA Egyptian patients, and their relationship to Methotrexate therapy, disease duration, and activity.

Patients and Methods: This was a cross sectional study which was done on 50 RA patients diagnosed according to Rheumatoid Arthritis - 2010 American college of rheumatology/ European League Against Rheumatism (ACR-EULAR) attending rheumatology and chest inpatient departments and outpatient clinics in Ain Shams University Hospitals.

Results: Patients were divided into two equal groups: Group A: - 25 RA patients treated with MTX only +/- low dose steroid. Group B: - 25 MTX naive RA patients (treated with DMARDs other than MTX) +/- low dose steroid.

Conclusion: We found MTX has no role in RA-ILD, there is no significant difference between MTX users and MTX naïve regarding spirometry and HR-CT.

DETAILED DESCRIPTION:
This was a cross-sectional study which was done on 50 RA patients diagnosed according to Rheumatoid Arthritis - 2010 American college of rheumatology/ European League Against Rheumatism (ACR-EULAR) classification criteria (Aletaha et al., 2010), patients enrolled from rheumatology and chest inpatient departments and outpatient clinics in Ain Shams University Hospitals.

Patients were divided in to two equal groups:

- Group A: - 25 RA patients treated with MTX only +/- low dose steroid

. Group B: - 25 MTX naive RA patients (treated with DMARDs other than MTX) +/- low dose steroid.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 yr rheumatoid arthritis more than one year, all patients were under RA Treatment for more than one year

Exclusion Criteria:

* Patients with recent respiratory infection, history of pulmonary tuberculosis or other chest disorders such as COPD, bronchial asthma, vasculitis, pleural diseases, thromboembolism or pulmonary hypertension, any patient receiving drugs that induce ILD such as chemotherapeutics, antimicrobials, cardiovascular agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 50 RA patients diagnosed according to Rheumatoid Arthritis - 2010 American college of rheumatology/ European League Against Rheumatism (ACR-EULAR) attending rheumatology and chest inpatient departments and outpatient clinics in Ain Shams University Hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
HRCT Chest and spirometry test findings in RA Egyptian patients, and their relationship to Methotrexate therapy, disease duration, and activity. | 7 months
  50 RA patients diagnosed according to Rheumatoid Arthritis - 2010 American college of rheumatology/ European League Against Rheumatism (ACR-EULAR) classification criteria (Aletaha et al., 2010), patients enrolled from rheumatology and chest inpatient departments and outpatient clinics in Ain Shams University Hospitals, and had spirometry, HRCT chest to assess methotrexate pulmonary afffection

CONTACTS AND LOCATIONS:
Overall Officials: Heba M Shalaby, MD, Principal Investigator — Ain Shams University, Faculty of medicine
Locations (1):
- Faculty of medicine, Ain Shams University, Cairo, Egypt